CLINICAL TRIAL: NCT05151120
Title: Harmonization of Thyroid-stimulating Hormone Immunoassays Reagents - Blood Collection From Patients With Thyroid Disorders
Brief Title: Harmonization of Thyroid-stimulating Hormone Immunoassays Reagents
Acronym: IFCC-TSH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0806; 2021-A02187-34 (Other: ID-RCB)
Record Dates: First submitted 2021-10-21; First posted 2021-12-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Disorders; Thyroid Stimulating; Hormone, C
Keywords: Blood Sample collection; TSH results harmonisation; IVD-manufacturers; Reference intervals; Results harmonisation
MeSH Terms: conditions — Thyroid Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 sample during routine venepuncture of 49 mL blood collection (7 x 7mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Hyperthyroid: 30 patients will be included and divided into three categories: A1: 10 patients with suppressed TSH, around 0.01 milli-international unit/liter (mIU/L) A2: 10 patients with TSH values between 0.01 - 0.1 mIU/L A3: 10 patients with TSH values between 0.1 - 0.4 mIU/L
  Interventions: Biological: blood sample
- Group B: Euthyroid: 30 Patients (under treatment) with TSH values between 0.4 - 4 mIU/L will be included
  Interventions: Biological: blood sample
- GROUP C: Hypothyroid: 40 patients will be included and divided into two categories: C1: 20 patients with TSH values between 4 - 50 mIU/L C2: 20 patients with TSH values > 50 mIU/L up to 100 mIU/L. Even distribution (if possible).
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — In practice the only intervention of the study is 49 mL extra blood along with the blood draw that is already planned for diagnosis/follow-up

SUMMARY:
Given the prevalence and gravity of thyroid disorders, timely diagnosis, initiation, and monitoring of therapy are important to restrict the impact of the disease on public health. Measurement of serum thyroid stimulating hormone (TSH) concentrations is an indispensable tool to confirm the disease and clinical management.

Reference intervals (RI) reported along with the laboratory data are an integral part of the interpretation process. Since many laboratory measurements are not yet comparable, RIs are typically established for each assay and are considered assay-specific. In this context, physicians who request test results from different laboratories are faced with challenges owing to different RIs. Assay-specific RIs are also problematic for patients who are seen by different doctors/different countries and more generally, assay-specific measurement results limit the development of modern public health standards.

Paramount to the goal of using common RIs is the establishment of metrological traceability of in vitro diagnostic (IVD) medical devices-also called standardization. As the International Federation of Clinical Chemistry (IFCC) Committee for Standardization of Thyroid Function Tests (C-STFT) members, the investigators decided to focus efforts on immunoassays for TSH in partnership with the IVD industry.

Although a reference measurement procedure existed for free thyroxine, the investigators considered this option for TSH unlikely and developed a pragmatic approach to harmonization rather than standardization.

Harmonization is important in order to guarantee comparability of results obtained in different laboratories. The harmonization process is conducted by assigning target values to a large set of samples, based on the results obtained by as many IVD-manufacturers as possible (ref 2). Important here is the fact that these samples must cover the full measuring range of a TSH assay, and so it is necessary to include samples from people with thyroid disease.

The primary objective of the study is the constitution of blood samples collection from patients with thyroid disorders in order to harmonize several commercially available immunoassays used for the determination of thyroid hormone concentrations in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Body weight ≥ 62 kg
* With a thyroid disorder (with high, low or normal TSH levels)
* Competent to give non opposition after information

Exclusion Criteria:

* Age <18 years old
* Those individuals previously enrolled into this clinical study
* Individuals diagnosed with a severe non-thyroidal illness at physician's appreciation. Defined as a state of dysregulation where levels of T3, T4, free triiodothyronine (FT3) and/or free thyroxine (FT4) are abnormal although the Thyroid gland does not appear to be dysfunctional. In practice, non-thyroidal illness (NTI) is reported to be usually associated with critical illness or starvation. Examples: chronic renal failure, liver cirrhosis, advanced (active) malignancy, sepsis, trauma, prolonged fasting or starvation, heart failure, Myocardial infarction (MI), and any psychiatric disorder.
* Pregnancy - please note that pregnancy test is not needed, a declaration is sufficient. The inclusion of a sample from a woman with an unidentified pregnancy will not jeopardize the study.
* Patient under guardianship and under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment will be performed from the clinical cohort of thyroid disorder patients followed at the Hospices Civils de Lyon Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Number of subjet included | through study completion, an average of 18 months
  The primary objective is to collect 100 blood samples that distributed into the followings groups:
  GROUP A: Hyperthyroid (N = 30) A1: 10 patients with suppressed TSH, around 0.01 mIU/L A2: 10 patients with TSH values between 0.01 - 0.1 mIU/L A3: 10 patients with TSH values between 0.1 - 0.4 mIU/L
  GROUP B: Euthyroid (N = 30) Patients (under treatment) with TSH values between 0.4 - 4 mIU/L
  GROUP C: Hypothyroid (N = 40) C1: 20 patients with TSH values between 4 - 50 mIU/L C2: 20 patients with TSH values > 50 mIU/L up to 100 mIU/L.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service D'endocrinologie - Hôpital Louis Pradel - Hospices Civils de Lyon, Bron
  - Service de Médecine Nucléaire - Hôpital Louis Pradel - Hospices Civils de Lyon, Bron